CLINICAL TRIAL: NCT07308210
Title: Developing a Home-based Executive Function Training Program for Autistic Individuals
Brief Title: Hybrid Computerized EF Training Using Virtual Human Stimuli for Autism
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Responsible Party: Principal Investigator, YEUNG Kin Chung Michael, Assistant Professor, Education University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-2023-0504
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid computerized executive function training (Experimental): Hybrid computerized executive function training five 30-minute sessions a week, for two weeks.
  Interventions: Behavioral: Hybrid computerized executive function training

INTERVENTIONS:
Behavioral: Hybrid computerized executive function training — The Face-Judgment game trains shifting through 33 trials where players judge a face's sex or emotion based on cues. Trials include repeat or switch judgments, with cue durations decrease from 1,000 ms to 200 ms to increase difficulty. Performance metrics include mean switch RT and switch cost RT for adjusting difficulty. The Gaze-Arrow game enhances inhibition by requiring players to process gaze direction amidst distractors. Each round has 32 trials with faces and arrows pointing left or right. Arrow pairs increase from 1 to 5 across levels, increasing interference in incongruent trials, where gaze and arrow directions mismatch. Players judge gaze direction; performance is measured by mean incongruent RT and interference score. The Running Memory game trains working memory by having players recall face identities from n trials earlier, with n increasing from 1 to 5. Afterward, players select the face matching the cue from five options, with accuracy guiding level adjustments.

SUMMARY:
The goal of this pilot clinical trial is to learn the preliminary feasibility and efficacy of a home-based hybrid computerized executive function (EF) training program using social stimuli for autistic individuals. The main questions it aims to answer are:

1. Does hybrid EF training using virtual human stimuli improve the EF and symptoms of autistic individuals?
2. What are the parents' attitudes toward the training program?

Researchers will compare changes in EF task performance and parent-report autistic symptoms and investigate parents' responses on a feedback questionnaire after autistic individuals undergo two weeks of training.

Participants will:

1. Undergo computerized training at home five 30-minute sessions a week, for two weeks
2. Visit the university campus before and after the training program to undertake an assessment

DETAILED DESCRIPTION:
To facilitate the integration of executive functioning (EF) and socio-emotional cue processing, we developed a novel home-based EF training program utilizing virtual, culturally relevant human facial stimuli for autistic individuals. We will ask autistic participants aged 8-17 to engage in training using this newly developed application at home over a two-week period, with five 30-minute sessions per week.

The newly developed hybrid computerized training application features three games targeting the three core components of executive function (EF): shifting, inhibition, and updating (Miyake et al., 2000). These games utilize 20 virtual Asian characters generated with Character Creator 4 (Reallusion Inc.).

The Face-Judgment Game (Categorization or "分門別類") trains shifting and mental flexibility by involving sex and emotion judgments (de Vries & Geurts, 2012). Each round has 33 trials. Trials begin with a blank period, followed by a cue period lasting between 2000 ms and a decreasing duration from 1000 ms to 200 ms as difficulty increases. The cue is either "Sex" or "Emotion." After these periods, a face displaying happiness or fear is shown at the center of the screen. The player judges the face's sex (male/female) or emotion (happy/scared) based on the cue, responding as quickly and accurately as possible. Trials are either repeat trials (same judgment as previous) or switch trials (different judgment). Performance indices include mean switch reaction time (RT) and switch cost RT, used for difficulty adjustment.

The Gaze-Arrow Game (Point Out The Way or "指點迷津") trains inhibition and interference control by requiring processing gaze direction amid distractors (Eriksen & Eriksen, 1974). Each round has 32 trials. Trials start with a blank period, then present a neutral or emotional face along with arrow flankers pointing left or right. The number of arrow pairs increases from one to five across levels, creating greater interference when target and flanker directions mismatch (Chanceaux et al., 2014). The player judges gaze direction. Trials are either congruent (gaze and arrows same direction) or incongruent (opposite directions). Performance is measured by the mean incongruent RT and the RT difference between incongruent and congruent trials (interference score), used for level adjustment.

The Running Memory Game (Character Memorization or "人物記憶") trains updating working memory by processing face identities (Morris & Jones, 1990). Each trial begins with an instruction cue, followed by a sequence of neutral or emotional faces. The cue prompts the player to remember a face from n trials earlier, with n increasing from 1 to 5 to impose greater working memory demands. The sequence length varies randomly from 6 to 10 faces, with no repeated identities. After the sequence, five recent faces are shown, and the player selects the face matching the cue. Accuracy serves as the performance index for level adjustment.

Assessments of participants' EF and clinical symptoms will be conducted within one week before the first training session and within one week after the last training session. Additionally, we will examine parents' attitudes toward the program.

The go/no-go task measures inhibition (Picton et al., 2007). It requires participants to press a button in response to one letter (go trials) and to withhold responses to other letters (no-go trials). Each trial consists of a letter appearing for 300 ms, followed by an interstimulus interval of 1,000 to 1,400 ms (mean = 1,200 ms). The go:no-go ratio is 3:1, with 240 go trials and 80 no-go trials. The false alarm rate is analyzed.

The Sternberg working memory task assesses the storage and retrieval of items from short-item memory (Sternberg, 1966). It requires participants to remember sets of 3 or 6 capital English letters, one by one. The two set sizes are equiprobable and presented in a randomized order. On each trial, participants see a fixation cross for 500 ms, followed by the letter stimuli presented for 2,000 ms. This is followed by a 3,000-ms blank period, then a lowercase letter probe appears for 1,000 ms, followed by an interstimulus interval of 1,750 to 2,250 ms (mean = 2,000 ms). The response time window is 2,750 ms. There are28 trials for each set size. Accuracy at set size 6 is analyzed.

The digit task-switching task measures shifting (Monsell, 2003). On each trial, a fixation cross is shown for 500 ms. Next, a cue indicating either "large/small" (magnitude judgment) or "odd/even" (parity judgment) is presented either at 0 ms or 1,000 ms before a single digit, ranging from 1 to 9 (excluding 5). Upon seeing the digit, participants are required to judge the digit according to the cue as fast as possible via a button press. A repeat trial occurs when the current judgment is the same as the previous one, and a switch trial is defined when the present judgment differed from the last one. These two trial types and the two cue-target intervals are equiprobable, with 32 trials for each combination. The reaction time (RT) switch cost (i.e., difference in mean RT between repeat and switch trials) at 0-ms cue-target interval, which allows no preparation, is analyzed.

The Social Responsiveness Scale-2 (SRS-2) has 65 items measuring the social function deficits associated with autism (e.g., "has difficulty relating to peers") (Constantino & Gruber, 2012). Each item is rated on a 4-point scale from "0" (never true) to "3" (almost always true). The questionnaire yields two DSM-V compatible subscale scores, including the Social Communication and Interaction (SCI) and Restricted Interests and Repetitive Behavior (RRB) scores. The raw scores of these two subscales are analyzed.

A feedback questionnaire is completed by parents to evaluate their attitudes toward the training program and to collect suggestions for game improvement. They rate six items on a 7-point Likert scale, from -3 to +3. These items include 'interestingness of the training games' (from very boring to very interesting), 'difficulty of the training games' (from too easy to too difficult), 'duration of the training games' (from too short to too long), 'perceived change in the child following training' (from very negative to very positive), 'satisfaction with the overall arrangement of the training' (from very dissatisfied to very satisfied), 'willingness to have the child join similar cognitive training in the future' (from very unwilling to very willing).

We hypothesize that both EF and clinical symptoms will improve due to enhanced integration of EF and social-cognitive processes. The hypothesis will be confirmed by conducting t-tests on the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Having met the DSM-V-TR criteria for autism spectrum disorder
* Age between 8 and 17 years
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Any neurological conditions
* Head injuries requiring hospitalization

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The Go/No-Go Task - The false alarm rate | Within one week before the first training session and within one week after the last training session
  The percentage of false alarms made on no-go trials
The Sternberg Working Memory Task - Accuracy at set size 6 | Within one week before the first training session and within one week after the last training session
  The percentage of probes recognized when arrays of 6 letters are to be remembered
The Digit Task-Switching Task - Reaction time (RT) switch cost | Within one week before the first training session and within one week after the last training session
  Difference in mean RT between repeat and switch trials
The Social Responsiveness Scale-2 (SRS-2) - Social Communication and Interaction (SCI) raw score | Within one week before the first training session and within one week after the last training session
  A parent-reported measure of social functioning deficits associated with autism
The Social Responsiveness Scale-2 (SRS-2) - Restricted Interests and Repetitive Behavior (RRB) raw score | Within one week before the first training session and within one week after the last training session
  A parent-reported measure of behavioral inflexibility associated with autism
Parents' Feedback Questionnaire - Score | Within one week after the last training session
  Parents' attitudes toward various statements regarding the training program, rated on a 7-point Likert scale (from -3 to +3)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Yeung, PhD, Principal Investigator — The Education University of Hong Kong
Locations (1):
- The Education University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Chanceaux M, Mathot S, Grainger J. Effects of number, complexity, and familiarity of flankers on crowded letter identification. J Vis. 2014 Nov 10;14(6):7. doi: 10.1167/14.6.7. PMID 25384390
- [Background] de Vries M, Geurts HM. Cognitive flexibility in ASD; task switching with emotional faces. J Autism Dev Disord. 2012 Dec;42(12):2558-68. doi: 10.1007/s10803-012-1512-1. PMID 22456815
- [Background] Eriksen, B. A., & Eriksen, C. W. (1974). Effects of noise letters upon the identification of a target letter in a nonsearch task. Perception & psychophysics, 16(1), 143-149. https://doi.org/10.3758/BF03203267
- [Background] Miyake A, Friedman NP, Emerson MJ, Witzki AH, Howerter A, Wager TD. The unity and diversity of executive functions and their contributions to complex "Frontal Lobe" tasks: a latent variable analysis. Cogn Psychol. 2000 Aug;41(1):49-100. doi: 10.1006/cogp.1999.0734. PMID 10945922
- [Background] Morris, N., & Jones, D. M. (1990). Memory updating in working memory: The role of the central executive. British journal of psychology, 81(2), 111-121. https://doi.org/10.1111/j.2044-8295.1990.tb02349.x
- [Background] Constantino, J. N., & Gruber, C. P. (2012). Social responsiveness scale, Second Edition (SRS-2). Torrance, CA: Western Psychological Services.
- [Background] Monsell S. Task switching. Trends Cogn Sci. 2003 Mar;7(3):134-140. doi: 10.1016/s1364-6613(03)00028-7. PMID 12639695
- [Background] Picton TW, Stuss DT, Alexander MP, Shallice T, Binns MA, Gillingham S. Effects of focal frontal lesions on response inhibition. Cereb Cortex. 2007 Apr;17(4):826-38. doi: 10.1093/cercor/bhk031. Epub 2006 May 12. PMID 16699079
- [Background] Sternberg S. High-speed scanning in human memory. Science. 1966 Aug 5;153(3736):652-4. doi: 10.1126/science.153.3736.652. PMID 5939936